CLINICAL TRIAL: NCT05414578
Title: The Nordic IBD Study Within Personalized Medicine - Diagnosing and Prediction Using Molecular Characterization of Inflammatory Bowel Disease: the NORDTREAT Prospective Cohort Study
Brief Title: NORDTREAT Prospective Study on Inflammatory Bowel Disease
Status: Recruiting | Type: Observational
Sponsor: University of Southern Denmark (Other)
Collaborators: Nordic Bioscience A/S (Industry); University Hospital Bispebjerg and Frederiksberg (Other); Aalborg University (Other); Colitis-Crohn Foreningen (Other); Uppsala University (Other); Örebro University, Sweden (Other); Lovisenberg Diakonale Hospital (Other); University of Oslo (Other); University of Kiel (Other); University Hospital of Southern Denmark (Unknown)
Responsible Party: Sponsor
Other Study IDs: NORDTREAT_MOK 2022
Record Dates: First submitted 2022-04-28; First posted 2022-06-10 (Actual); Last update posted 2022-06-10 (Actual); Status verified 2022-06

CONDITIONS: Inflammatory Bowel Diseases (IBD); Crohn Disease (CD); Ulcerative Colitis (UC)
Keywords: Prospective clinical study; Biomarkers; Diagnosis; Prognosis
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 52 Weeks
Biospecimen Retention: Samples With DNA — Intestinal biopsies, blood, urine, feces and hair
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Inflammatory bowel disease (IBD), primarily ulcerative colitis (UC) and Crohn's disease (CD), is a chronic disease entity affecting individuals of all ages, and which may severely impact the lives of the patients and their families as well as society. Individuals with IBD may have to live with relapsing symptoms, such as diarrhea, abdominal pain, and fatigue. Further, a substantial proportion of patients develop serious complications such as bowel obstruction and fistula, and some develop complicating liver disease and eventually colorectal cancer. The consequences are that many patients suffer hospitalizations, recurring sick-leave, life-long medication, and surgical interventions. As IBD has become increasingly common in Western populations there is a clear need to improve the outcome from IBD.

IBD is a heterogeneous disease entity with substantial differences between patients and personalized medicine may help provide strategies for better treatment . Currently, one of the main unmet needs is the glaring lack of robust biomarkers for individual disease characterization. This lack leads to delayed diagnosis, worse outcomes, increased mortality and an amplified disease burden. Furthermore, diagnosis of IBD is difficult and early diagnosis is crucial as it helps avoid the development of irreversible organ damage. Therefore, there is an emerging focus on the development of simple, non-invasive, and cheap biomarkers to support clinical decision-making in IBD.

This Nordic, prospective, clinical study has the aim of identifying markers that are associated with the diagnosis of IBD and prediction of clinical outcomes with various disease manifestations. Importantly, this study will evaluate the markers in a relevant clinical setting, i.e. among patients referred to the hospital for suspicion on IBD using the ECCO Criteria.

Specifically the aims of the study are to:

* Improve the accuracy to diagnose IBD
* Improve the accuracy to define the prognosis of IBD

The study is approved by the local Ethics Committee (S-20200051) and the local Data Agency (20/54594).

DETAILED DESCRIPTION:
The primary aim is to identify molecular markers (e.g. in the blood and stools) for discrimination between individuals diagnosed with inflammatory bowel disease (IBD) inclusive Crohn's disease (CD), ulcerative colitis (UC) and inflammatory bowel disease unclassified (IBD-U), and those without (non-IBD). Participants with suspected IBD at baseline, with various disease pathways, will be evaluated again using a 1-year cohort study. Diagnosis and clinical outcome will be evaluated at referral and after 1 year of observation.

The secondary aims are, in addition to the molecular information, to investigate whether the inclusion of information on clinical and lifestyle factors as well as combination hereof (e.g. gene-environment interaction analyses) can improve the predictive potential of identifying IBD and distinguish the prognosis.

Study design: A prospective Nordic multicenter study on prognostic factors for the diagnosis and characterization of IBD among patients referred to the hospital on suspicion of IBD. A panel of possible prognostic biomarkers for diagnostic purposes will be applied to all participants.

Setting: All patients referred due to a suspicion of IBD to the departments of gastroenterology in Odense University Hospital, Svendborg Hospital, Vejle Hospital, Esbjerg Hospital and potentially Hospital of Southern Jutland, Aabenraa will be invited to take part in the study. Participants will be included from January 2022 for a 1-year period or until 800 participants in the Nordic study (up to 400 in Denmark) have been included. The follow-up period is one-year including visits and questionnaires and an additional nine years of follow-up by the use of register data. Biological material will be obtained four times for participants with IBD, at week-2/0, and 12, 26 and 52 after the diagnosis has been established. Participants where IBD is not established (non-IBD) will only have biological material obtained at baseline (that is visit -2/0) and will have a clinical interview after 52 weeks. All participants are treated according to standard clinical practice by the clinical departments.

Clinical data consist of personal data, data on health and disease, lifestyle, laboratory measures, and disease activity scores including patient-reported outcome measures (PROMs), clinical assessments, and laboratory data. Each participant will fill out validated questionnaires on disease activity, quality of life, and lifestyle using electronic links.

Data management: Study data registered by clinicians, study nurses and technicians will be stored in the web-based case report form (eCRF) Viedoc (Viedoc™, Uppsala, Sweden) or REDCap (Open Patient data Explorative Network (OPEN) at Odense University Hospital) for the diet questionnaire. The questionnaires are in Danish and the participants will have access to the questionnaires via an electronic link sent to their personal, electronic mailbox (REDCap) or via an investigator provided link to MyViedoc. All data will be stored in secure research storage facilities.

Statistical methods: We will develop multivariable prediction models relating multiple predictors for a particular individual to the probability of or risk for the presence (diagnosis of IBD at baseline) or future occurrence (prognosis) of a particular outcome such as severe IBD within the first year. Predictors such as biomarkers are covariates, explored as prognostic factors (independent variables).

The primary hypothesis is that the final biomarker will define the participant population into two groups each consisting of 50%: a biomarker positive group whereof 80% will be diagnosed with IBD and a biomarker negative group whereof 20% will be diagnosed with IBD.

For a comparison of two independent binomial proportions using the likelihood ratio statistic with a Chi-square approximation with a two-sided significance level of 0.05, a total sample size of 800 assuming a ratio biomarker positivity-to-negativity of 1 to 1 has an approximate power of 100% when the proportions of being diagnosed with IBD are 0.8 and 0.2. If we assume that we will have 800 study participants, we will potentially ("rule of thumb") be able to build a statistical model with as many as 80 covariates in the multivariable model.

The associations of the suspected important biomarkers with other variables will be tested with non-parametric tests: with Spearman rank correlation (rs) for continuous variables, and the Wilcoxon rank-sum test or Kruskal-Wallis test, including a Wilcoxon-type test for trend across ordered groups where appropriate, for categorical variables. In general, logistic regression models will be used with individual marker as the exposure variables and the clinical response as the outcome (dependent variable). The analyses will be adjusted simultaneously for sex, age, and prescribed targeted therapy. Potential interaction between biomarker status (positive/negative) and specific drug type will be analyzed. Covariates (biomarkers) consist of various measures within genetics, transcriptomic, microbiomes, and proteomics.

Sample size considerations: Assuming that biomarker positivity constitutes 50% of the individuals enrolled at baseline, if our event rate is 10% on average, a total sample size of 800 patients (i.e. 400 biomarker positive) we will have a very good statistical power (99.7%) to detect a difference between proportions having surgery of 10% points (15% and 5%, respectively). If we decide to split the data set into two (2×400 individuals), in order to first build the model, and subsequently validate it in the second independent dataset, we will have 91.8% statistical power to detect a difference between groups. If the prognostic value of our biomarkers is not that effective separating the number of patients with severe IBD at week 52, we will still have more than 90% power to detect a difference between biomarker groups of 6% points (e.g. 10% and 4%, respectively).

Another consideration is the number of events (individuals having severe IBD at week 52) per variable (EPV) considered for inclusion in the multivariable model. For logistic regression modelling the EPV should be at least ten times the number of potential prognostic variables that could be included in the model. As a consequence of this logic, our expected sample size of 800 individuals (having 80 events) will, with reasonable confidence, allow us to create a multivariable model with up to 8 covariates simultaneously.

Project organization: NORDTREAT is part of a larger Nordic project (DK, SE, NO and IS) where regular meetings will be held between the partners. Collaborative research and material transfer agreements will be conducted with the national and international collaborators.

In addition to the scientific reporting of results, major findings with translational implications will be communicated to health professionals, patient organizations, public health policy makers, and to the general public through various media and news activities.

ELIGIBILITY:
To be included in the study, the participants must meet the following criteria:

Inclusion Criteria:

* Referred on the suspicion of inflammatory bowel disease
* Adult (+18 years of age)
* Written informed consent to participate in the study

Exclusion Criteria:

* A previous known diagnosis of Crohn's disease, ulcerative colitis or IBD-U
* Unable to provide informed consent
* Unable to comply with protocol requirements (e.g., for reasons including alcohol and/or recreational drug abuse)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred to the hospital on suspicion of IBD
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2022-02-07 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2031-01 (Estimated)

PRIMARY OUTCOMES:
Improving the accuracy to diagnose IBD | Baseline (Week 0) and Week 52
  The primary endpoint in the cross-sectional study will be diagnosis, i.e., IBD (including CD, UC, IBD-U) or non-IBD (patients that are not diagnosed with IBD) at referral. IBD is diagnosed according to the ECCO criteria based on endoscopic, histologic and/or radiological criteria.
Improving the accuracy to define prognosis of IBD | Week 52
  The primary endpoint in the longitudinal cohort study will be severe IBD at week 52 defined as:
  * IBD-related surgery or
  * IBD-related hospitalization (except planned procedures) or
  * IBD-related death

SECONDARY OUTCOMES:
Lack of corticosteroid-free clinical remission at week 12* | Week 12
  ● Clinical remission, CD: Patient reported outcome 2 (abdominal pain ≤ 1 and stool frequency ≤ 3) or Harvey Bradshaw Index < 5
  ● Clinical remission, UC: Patient reported outcome 2 (rectal bleeding = 0 and stool frequency = 0) or Partial Mayo (< 3 and no score >1)
  *Both local acting systemic administered (budesonide) and systemic steroids (prednisolon)
Lack of corticosteroid-free endoscopic healing at week 52* | Week 52
  ● Endoscopic healing, CD: Simple endoscopic score in CD < 3 points or absence of ulcerations (e.g. SES-CD ulceration subscores = 0)
  ● Endoscopic healing, UC: Mayo endoscopic subscore = 0 points, or UC endoscopic index of severity ≤ 1 points
  *Both local acting systemic administered (budesonide) and systemic steroids (prednisolon)
Disease impact on patients life (daily functioning and quality of life) | Week 52
  ● The Inflammatory Bowel Disease Questionnaire (with a scale from 1-7); where
  1 is eg. "All of the time" and 7 is "At no time" or 1 is "No energy" and 7 is "Full of energy"
Disease impact on patients life (perception of health) | Week 52
  ● Short Form 36 is an 11-item questionnaire on the patient's perception of his/her health (with scales from 1-3, 1-5, 1-6 or yes / no) where e.g. 1 denotes "Excellent" and 5 denotes "Bad" or 1 denotes "No pain" and 6 denotes "Very strong pain".
Disease impact on patients life | Week 52
  ● The 14-item version of the IBD Disability Index (modified to be suitable as a self-report) is a questionnaire on IBD and perception of health. The scales range from eg.:
  * Very good / Good / Moderate / Bad / Very bad
  * Yes / No
  * None / Mild / Moderate / Severe / Extreme
Disease impact on patients life (fecal incontinence) | Week 52
  ● Fecal incontinence according to the Wexner score (with a scale from 0-20); where 0 is perfect continence and 20 is complete incontinence.
Mid-term complications | Week 52
  * Bowel damage in CD according to the Lémann index
  * IBD-related surgery and hospitalizations defined as:
    * Surgery, UC: any colectomy
    * Surgery, CD: any CD-related surgery
    * Hospitalizations: A composite endpoint combining the total number of IBD-related hospitalizations (including readmissions), and the cumulative length of hospital stay.
    * Disease extension in UC: focus on macroscopic proximal disease extension
Long-term complications | Week 52
  * Gastrointestinal and extra-intestinal dysplasia
  * Cancer
  * Mortality
Surgery in CD due to obstructive symptoms (stenosis) | Week 52
  Cumulative number of surgeries in CD due to stenosis
Anxiety and depression | Week 52
  Hospital Anxiety and Depression Scale (HADS) is a 14-item scale with seven items each for anxiety and depression subscales. Scoring ranges from 0 to 3 and a score above 8 denotes anxiety or depression respectively.
Fatigue Questionnaire | Week 52
  The Inflammatory Bowel Disease-Fatigue (IBD-F) Part One is a 5-item scale where scoring ranges from 0 to 4. Zero denotes no fatigue and 4 denotes extreme fatigue.
Flares | Week 52
  Cumulative number of flares at 1 year
Glucocorticoid exposures | Week 52
  Cumulative glucocorticoid exposures at 1 year
Adverse drug reactions | Week 52
  Cumulative number of adverse drug reactions
Increased faecal calprotectin at week 52 | Week 52
  Increased faecal calprotectin is defined as cumulative number of patients with a concentration of faecal calprotectin higher than 250 μg/g
Time to start of biological therapy | Week 52
  Cumulative number of days before start of biological therapy
Time to onset of event (IBD-related surgery or IBD-related hospitalization) | Week 52
  Cumulative number of days before onset of IBD-related surgery or IBD-related hospitalization
The composite secondary outcome of the proportion of patients who experience severe IBD within 52 weeks after inclusion | Week 52
  Cumulative number of patients who experience:
  * Need for medication between diagnosis and one year (immunomodulators, biologicals, steroids) or
  * Need for surgery between diagnosis and one year or
  * Need for hospitalization between diagnosis and one year or
  * Number of relapses between diagnosis and one year.

CONTACTS AND LOCATIONS:
Overall Officials: Jens Kjeldsen, Professor, Principal Investigator — Odense University Hospital; Vibeke Andersen, Professor, Principal Investigator — University Hospital of Southern Denmark, Aabenraa
Locations (17):
- Denmark (5):
  - University Hospital of Southern Denmark, Aabenraa
  - SVS Esbjerg Hospital, Esbjerg
  - Odense University Hospital, Odense
  - OUH Svendborg Hospital, Svendborg
  - SLB Vejle Hospital, Vejle
- Landspitali, Reykjavik, Iceland
- Norway (5):
  - Vestre Viken HF, Drammen
  - Østfold Kalnes, Grålum
  - Oslo Universitetssykehus, Oslo
  - Sykehuset i Telemark, Skien
  - Sykehuset i Vestfold, Tønsberg
- Sweden (6):
  - Höglandssjukhuset Eksjö, Eksjö, Region Jönköpings Län
  - Karolinska Universitetssjukhuset, Stockholm, Region Stockholm
  - Akademiska Sjukhuset Uppsala, Uppsala, Region Uppsala
  - Universitetssjukhuset i Linköping, Linköping, Region Östergötland
  - Ersta Sjukhus, Stockholm
  - Universitetssjukhuset Örebro, Örebro, Örebro County

REFERENCES:
- [Derived] Fejrskov A, Fuchtbauer JD, Daviethsdottir LG, Halfvarson J, Hoivik ML, Jensen MD, Mortensen JH, Nielsen LN, Rejler M, Repsilber D, Soderholm JD, Aalykke C, Andersen V, Christensen R, Kjeldsen J. Novel biomarker profiles to improve individual diagnosis and prognosis in patients with suspected inflammatory bowel disease: protocol for the Nordic inception cohort study (NORDTREAT). BMJ Open. 2024 May 15;14(5):e083144. doi: 10.1136/bmjopen-2023-083144. PMID 38754881